CLINICAL TRIAL: NCT05162118
Title: Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of VG161 in Combination With Nivolumab in Patients With Advanced Pancreatic Cancer
Brief Title: Clinical Study of VG161 in Combination With Nivolumab in Subjects With Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Chief of hepatobiliary and pancreatic surgical department, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VG161-IIS-201
Record Dates: First submitted 2021-11-23; First posted 2021-12-17 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Solid Tumor
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 1. Intratumoral injection of VG161 - 1.5*10^8 on D1 + Nivolumab on D8, D22
  2. Intratumoral injection of VG161 - 1.0*10^8 on D1, D2 + Nivolumab on D8, D22
  3. Intratumoral injection of VG161 - 1.0*10^8 on D1, D2, D3 + Nivolumab on D8, D22
  Interventions: Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) in combination with Nivolumab

INTERVENTIONS:
Drug: Recombinant Human IL12/15-PDL1B Oncolytic HSV-1 Injection (Vero Cell)) in combination with Nivolumab — Intratumoral injection of VG161 on day 1 only or day 1 through 3, in combination of Nivolumab intravenous injection only, Once every 2 weeks, 3 mg/kg each time.
  Other Names: VG161 + Nivolumab

SUMMARY:
VG161 is a recombinant human-IL12/15/PDL1B oncolytic HSV-1 Injectable. This is a multicenter, open, single-arm design clinical trial coducted in HSV-seropositive subjects with advanced pancreatic cancer to determine the safety, tolerability and preliminary efficacy of VG161 combined with PD-1 inhibitor (Nivolumab Injection).

DETAILED DESCRIPTION:
A multicenter, open, single-arm design of clinical trial of VG161 in combined with PD-1 inhibitor (Nivolumab) in the treatment of patients with advanced pancreatic cancer with metastasis. The standard 3 + 3 design was used in the dose-finding study to explore the safety of the combination treatment, determine the recommended safe dose (RP2D) of the combination treatment in the second phase of efficacy study. The first cycle was observed until Day 28, i.e., DLT observation period. In the efficacy investigation trial, Simon two-segment design was used to continue to investigate the preliminary efficacy of the combination at a safe dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give informed consent to this study before the trial and voluntarily sign a written informed consent form
* Age 18 to 75 years (inclusive), male or female
* According to the Guidelines for the Diagnosis and Treatment of Pancreatic Cancer, patients with histologically or cytologically confirmed advanced primary pancreatic ductal adenocarcinoma, acinar cell carcinoma or adenosquamous carcinoma, accompanied by metastasis (TxNxM1), who have failed standard treatment, or have no effective treatment at this stage
* The presence of at least one intratumoral injection lesion with the longest diameter (the longest diameter of lymph nodes) greater than or equal to 1.5 cm that is required by the dose volume of the acceptable current dose group, including superficial lesions or deep lesions that can be injected under B ultrasound/CT guidance (such as liver metastases, etc.)
* Herpes simplex virus type I (HSV-1) antibody test results (HSV-1IgG or HSV-1IgM) are positive
* ECOG performance score 0-1
* The expected survival time is more than 3 months
* Adequate organ function: 1) blood routine (No blood transfusion or colony-stimulating factor treatment Within 14 days): ANC ≥ 1.5 × 10^9/L, PLT ≥ 75 × 10^9/L, Hb ≥ 90 g/L, lymphocyte count ≥ 1.5 × 10^9/L (for lymphocyte count 1.0 × 10^9/L to 1.5 × 10^9/L, the investigator judges whether it is necessary); 2) liver function: TBIL ≤ 1.5 × ULN, ALT ≤ 3 × ULN, AST ≤ 3 × ULN (patients with liver metastases can receive ALT ≤ 5 × ULN, AST ≤ 5 × ULN); 3) Child-Pugh score: A-B; 4) renal function: Cr ≤ 1.5 × ULN, and creatinine clearance ≥ 45ml/min (calculated according to CockftGault formula); 5) coagulation function: activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 1.5 × ULN
* Eligible patients of childbearing potential (male and female) must agree to use a reliable method of contraception (hormonal or barrier method or abstinence) during the trial and for at least 90 days after medication; female patients of childbearing age must have a negative blood pregnancy test 7 days before inclusion

Exclusion Criteria:

* Received chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy (including PD-1/PD-L1 inhibitors) and other anti-tumor drug therapy 4 weeks before the first use of the study drug, oral fluoropyrimidines and small molecule targeted drugs are 2 weeks before the first use of the study drug or within 5 half-lives of the drug (whichever is longer)
* Received other unmarketed clinical trial treatment 4 times before the first use of the study drug
* Major organ surgery (excluding needle biopsy) or significant trauma 4 times before the first use of study drugs; 4. Patients who have received systemic corticosteroids (prednisone > 10 mg/day or equivalent doses of the same class of drugs) or other immunosuppressive agents within 14 days before the first use of study drugs; except for the following conditions: the use of topical, ocular, intra-articular, intranasal and inhaled corticosteroids; short-term use of corticosteroids for prophylaxis (such as prevention of contrast agent allergy)
* Have received vaccination 4 times before the first use of the study drug
* The adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except alopecia and other toxicities that are judged by the investigator to have no safety risk)
* Patients with central nervous system or spinal cord malignant tumors or metastases, which are not suitable for enrollment as judged by the investigator
* Accompanied by spinal cord compression, which is not suitable for the investigator's judgment
* In the period of herpes simplex virus recurrence and infection, and there are corresponding clinical manifestations, such as oral herpes labialis, herpetic keratitis, herpetic dermatitis, genital herpes and so on. 10.Other active uncontrolled infection
* History of immunodeficiency, including a positive HIV antibody test
* Patients with active hepatitis B or active hepatitis C. (Patients with hepatitis B virus carriers, stable hepatitis B after drug treatment [HBV-DNA negative] and cured hepatitis C [HCV RNA test negative]) were excluded. 13.History of severe cardiovascular disease: 1) arrhythmia requiring clinical intervention; 2) QTc interval > 480 ms; 3) acute coronary syndrome, congestive heart failure, stroke or other grade III and above cardiovascular events within 6 months; 4) New York Heart Association (NYHA) functional classification ≥ II or LVEF < 40%; 5) uncontrolled hypertension (judged by the investigator)
* Patients with active or previous autoimmune diseases that may relapse (such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); patients with clinically stable autoimmune thyroiditis, autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone, type I diabetes mellitus treated with stable doses of insulin, vitiligo or recovered childhood asthma/allergy, who do not require any intervention in adulthood
* Had received immunotherapy and experienced an irAE grade ≥ 3
* Known alcohol or drug dependence
* Patients with mental disorders or poor compliance
* Women who are pregnant or breastfeeding
* The subject has other serious systemic diseases or other reasons that make the subject unsuitable for this clinical study in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2022-03-08 (Estimated); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
MTD | 1 month
  MTD (Maximum tolerable dose)
Occurrence and numbers of DLT (phase 1) | 1 month
  Occurence of DLT (Dose Limiting Toxicity) and numbers of DLT
Occurence and frequence of AE and SAE (phase 1) | 24 month
  Occurence and frequence of Adverse Event (AE) and Serious Adverse Event (SAE) (NCI CTCAE 5.0)
DCR (phase 2) | 24 month
  Evaluate Disease Control Rate by RECIST 1.1
RP2D (phase 1) | 1 month
  RP2D (Recommended dose for phase II)

SECONDARY OUTCOMES:
DCR (phase 1) | 24 month
  Evaluate Disease Control Rate by RECIST 1.1
ORR | 24 month
  Evaluate Objective Response Rate by RECIST 1.1
PFS | 24 month
  Evaluate Progression Free Survival by RECIST 1.1
PD-1 | 24 month
  PD-1 level in peripheral blood T cells
Single cell sequencing | 24 month
  Single-cell sequencing of tumor biopsy samples
Occurence and frequence of AE and SAE (phase 2) | 24 month
  Occurence and frequence of Adverse Event (AE) and Serious Adverse Event (SAE) (NCI CTCAE 5.0)
CD3+ | 24 month
  Concentration of CD3+
CD4+ | 24 month
  Concentration of CD4+
CD8+ | 24 month
  Concentration of CD8+
CD4+/CD8+ | 24 month
  Concentration of CD4+/CD8+
NK | 24 month
  Concentration of NK
CD19+ | 24 month
  Concentration of CD19+
CD56+ | 24 month
  Concentration of CD56+
IL-6 | 24 month
  Cytokine levels of IL-6
TNF-a | 24 month
  Cytokine levels of TNF-a
IFN-γ | 24 month
  Cytokine levels of IFN-γ
CA19-9 | 24 month
  Tumor markers of CA19-9
CA125 | 24 month
  Tumor markers of CA125
CEA | 24 month
  Tumor markers of CEA

CONTACTS AND LOCATIONS:
Overall Officials: Tingbo Liang, Doctor, Principal Investigator — The First Affiliated Hospital Zhengjiang University School of Medicine
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No